CLINICAL TRIAL: NCT02262819
Title: Human Immunity Against Staphylococcus Aureus Skin Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 140199; 14-I-0199
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2019-04-24

CONDITIONS: Staphylococcus Aureus Skin Infection
Keywords: Skin Blister; Immune Response; Suction Device; Anti-Microbial; Killed Microbe
MeSH Terms: conditions — Blister

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: S. aureus — S. aureus, commensal coagulase-negative staphylococcal species, and Gram-negative commensals, such as Roseomonas and Pseudomonas species

SUMMARY:
Background:

- Staphylococcus aureus, or staph, is commonly found on the skin and in the respiratory system. Sometimes people who get sick with staph infection do not get better with standard treatment. These staph infections can be serious and even deadly. Researchers want to find out why some people are more likely to get the infection.

Objectives:

- To look at the immune response of the skin when it is exposed to bacteria.

Eligibility:

* People age 2 65 with hyper IgE syndrome (HIES) and those with recurrent staph infections.
* Healthy volunteers.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Over 1 5 days, participants may have blood tests and a skin and nasal swab. They may have additional tests if needed. If they had a recent biopsy, researchers may ask for a sample from it.
* Some participants will spend the night at the clinic. Their vital signs will be taken and they will have blood drawn. Some participants will take aspirin or ibuprofen starting 2 days before their stay.
* Some participants will have blisters created on the inside of their forearm. Suction will pull a layer of skin from their arm. Skin will be removed. Different solutions will be applied to the blisters. Up to 3 biopsies may be taken.
* Children will not have blood tests or biopsies.
* Participants will be called every day for 10 days, then at 30 days after the procedure.
* Participants will have a follow-up visit 10 days after the procedure.
* Participants who did not get blisters or biopsies will not have any follow-up appointments.

DETAILED DESCRIPTION:
The incidence of community-associated (CA) staphylococcal infections, especially those caused by methicillin-resistant Staphylococcus aureus (MRSA), has increased dramatically in recent years. Skin and soft tissues are the primary site for most of these infections, and skin or mucosal colonization increases the risk of disseminated disease. Many patients without apparent underlying immune dysfunction suffer from recurrent and persistent skin infections with MRSA. Additionally, patients with conditions such as atopic dermatitis and Hyper IgE (or Job s) Syndrome (HIES) are disproportionately affected. Although underlying host molecular defects responsible for some of these predisposing conditions have been uncovered in recent years (e.g. STAT3 mutations in HIES), the skin immune response to S. aureus infections has not been elucidated in either healthy controls or susceptible populations. In this protocol, we will perform exploratory evaluations of anti-staphylococcal immune responses in healthy subjects, subjects with STAT3 mutations, and otherwise healthy subjects with a history of recurrent staphylococcal skin infections. An additional group of subjects with other underlying conditions of interest may be included.

The primary objective of this research is to perform in vivo and ex vivo challenges with killed bacteria through the use of the skin blister model and keratinocyte cultures to evaluate skin immune responses. Occasionally, a commensal fungi, such as Candida species may also be used. We will use three experimental approaches to complete this objective: 1) evaluation of in vivo responses in skin blisters to killed microbe exposure, 2) ex vivo evaluation of anti-microbial responses through derivation of keratinocyte cultures from skin blisters or biopsies, and 3) evaluation of function and immune-stimulatory ability of commensal organisms.

Specifically, a suction blister device will be used to induce a skin blister on the forearm. The tops of the blisters will be removed, and solutions of killed S. aureus, commensal coagulase-negative staphylococcal species, or other Gram-negative commensals as well as commensal fungi, such as Candida species will be applied to the blisters to stimulate inflammatory responses. The blister fluid will then be collected at various time points over 24 hours for laboratory analysis. Baseline skin and/or nasal swabs, skin biopsies, and blood draws will also be performed (The skin and nasal swabs may be performed at the screening or baseline visit.). Pediatric participants may be enrolled for baseline skin and/or nasal swabs. All research procedures will be performed at the National Institutes of Health Clinical Center. We anticipate that the research will provide critical new information on the human skin immune response to S. aureus that has direct relevance for the development of vaccines, diagnostics, and therapeutics.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must either:

1. Have documentation of a proven or suspected immune defect or a history of invasive infection or recurrent (2 or more) skin infections with S. aureus (patient population); or
2. Not have evidence of an immune defect or history of invasive or recurrent S. aureus infections (healthy volunteers).

   * Participants must be between 2 and 65 years old (inclusive).
   * Participants must be willing to allow storage of blood, DNA, RNA, bacterial and fungal cultures, and other tissue samples for future research. Some research blood may not be required of healthy volunteers, except at the discretion of the Principal Investigator (PI).

EXCLUSION CRITERIA:

The following exclusion criteria apply to all participants:

* Current chemotherapy or underlying malignancy.
* Current oral steroids.
* Individuals with any condition that, in the opinion of the investigator, contraindicates participation in the study will be excluded.

The following exclusion criteria apply to adult participants in the blister portion of the study (Arm 1) only:

* Viral hepatitis B or C. Test results, including those from an outside facility or lab, within the prior 6 months will be accepted.
* HIV positive. Test results, including those from an outside facility or lab, within the prior 6 months will be accepted.
* Individuals on anticoagulant or anti-platelet therapy (other than aspirin or NSAIDs as described in the protocol).
* Pregnancy.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-10-10; Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the local in vivo skin immune response to bacteria. | 4 years
Evaluate the keratinocyte responses to bacterial challenge. | 4 years

SECONDARY OUTCOMES:
Determine if abnormalities in specific immune pathways, such as IL-17 and vitamin D metabolism, are present in subjects with recognized susceptibility to S. aureus infections. | 4 years
Characterize cultured skin bacteria (S. aureus, S. epidermidis, and other skin commensals) with molecular and functional studies. | 4 years
Assess the impact of non-steroidal anti-inflammatory drugs (NSAIDs) on skin immune function. | 4 years
Characterize blood immune parameters in a cohort of patients with invasive and/or recurrent skin and soft tissue S. aureus infections. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gough P, Ganesan S, Datta SK. IL-20 Signaling in Activated Human Neutrophils Inhibits Neutrophil Migration and Function. J Immunol. 2017 Jun 1;198(11):4373-4382. doi: 10.4049/jimmunol.1700253. Epub 2017 Apr 19. PMID 28424238
- [Background] Sastalla I, Williams KW, Anderson ED, Myles IA, Reckhow JD, Espinoza-Moraga M, Freeman AF, Datta SK. Molecular Typing of Staphylococcus aureus Isolated from Patients with Autosomal Dominant Hyper IgE Syndrome. Pathogens. 2017 Jun 6;6(2):23. doi: 10.3390/pathogens6020023. PMID 28587312